CLINICAL TRIAL: NCT04587089
Title: Efficacy of Guedes-Pinto Paste and CTZ Paste in the Non-instrumental Endodontic Treatment of Primary Teeth - Study Protocol for a Randomized Controlled Clinical Trial
Brief Title: Efficacy of Guedes-Pinto Paste and CTZ Paste in the Non-instrumental Endodontic Treatment of Primary Teeth
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Collaborators: Universidade Metropolitana de Santos (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EndoDeciduos
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Necrotic Pulp
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The clinical, radiographic and microbiological evaluations will be made by an assessor who will not know to which group the participants belong.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-instrumental Endodontic Treatment (NIET) + Guedes-Pinto Paste Group (Experimental): In this group, the canals will not be instrumented and the filling will be performed with Guedes-Pinto paste.
  Interventions: Procedure: Irrigation; Procedure: Filling with Guedes-Pinto Paste
- Non-instrumental Endodontic Treatment (NIET) + CTZ Paste Group (Experimental): In this group, the canals will not be instrumented and the filling will be performed with CTZ paste (Chlorophenicol, Tetracycline and Zinc Oxide and Eugenol).
  Interventions: Procedure: Irrigation; Procedure: Filling with CTZ Paste

INTERVENTIONS:
Procedure: Irrigation — Irrigation and aspiration in the root canals with 1% sodium hypochlorite (Milton's solution).
Procedure: Filling with Guedes-Pinto Paste — The root canals will be filled with Guedes-Pinto Paste, which is a composite of 3 medications: Rifocort® (dermatologic ointment), camphorated paramonochlorophenol (PMCC) and iodoform. It will be prepared at the moment of use with the same proportion in volume of 3 visually identical parts, one for each of its components.
  Arms: Non-instrumental Endodontic Treatment (NIET) + Guedes-Pinto Paste Group
Procedure: Filling with CTZ Paste — The powder that composes the CTZ paste will be previously manipulated in a 1:1:2 ratio (500mg of Chloramphenicol, 500mg of Tetracycline and 1,000mg of Zinc Oxide) by Formula & Ação (F&A) and incorporated into the eugenol liquid at the time of use, with the aid of a flexible spatula nº 24 and on a sterile glass plate. The cleaning of the coronary chamber must be carried out with saline solution and drying with sterile cotton balls and the CTZ paste must be inserted into the cavity.
  Arms: Non-instrumental Endodontic Treatment (NIET) + CTZ Paste Group

SUMMARY:
The maintenance of the deciduous tooth until its physiological exfoliation occurs is one of the main objectives of pediatric dentistry. Endodontic treatment in deciduous teeth resulting from carious or traumatic lesions with pulpal involvement is often necessary and we often find it difficult to perform it, due to the difficult control of the child, the internal anatomy of the root canals, and root resorptions. The non-instrumental endodontic treatment technique (TENI) associated with antimicrobial drugs has advantages such as shorter chair time and less complexity than the conventional technique in which root canal instrumentation is performed. The objective of this study is to carry out a controlled and randomized clinical trial to compare the effectiveness of non-instrumental endodontic treatment (NIET) in primary teeth associated with the use of two filling pastes. 120 necrotic deciduous teeth of children aged between 3 and 6 years will be selected; and the teeth will be divided into two groups. In Group 1 and Group 2, the root canals will not be instrumented, just irrigated and filled with the respective pastes, CTZ and Guedes-Pinto. The radiographic aspects will be evaluated, considering the repair process, clinically will be evaluated: presence of fistula and mobility, the evaluations will be carried out in both groups on the day of treatment and in periods of 1, 3 and 6 months after treatment. The data obtained will be submitted to the Shapiro-Wilk normality test, where the statistical analysis that will be used for this study will be defined, adopting a significance level of 95% (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3 to 6 years old with at least one anterior deciduous tooth with pulp necrosis in a position to be restored and at least 2/3 of the remaining root.
* Healthy patients and who did not antibiotic treatment in the previous three months.

Exclusion Criteria:

• Compromised health, primary teeth with more than one third root loss, lack of internal pathological resorption, impossibility of restoration, cases of re-treatment and crypt involvement.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-08-20 (Estimated); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Clinical Investigation of the Change in the Presence of Fistulas in Each Treated Tooth | Baseline, one month, 3 months and 6 months after treatment.
  In the follow-up consultations, teeth and gums will be clinically evaluated to check the presence of fistulas.
Clinical Investigation of Changes in Tooth Mobility in Each Treated Tooth | Baseline, one month, 3 months and 6 months after treatment.
  In the follow-up consultations, teeth will be clinically evaluated to check the presence of mobility.

SECONDARY OUTCOMES:
Radiographic Evaluation of the Changes in the Presence of Periapical Lesions in Each Treated Tooth | One month, 3 months and 6 months after treatment.
  In the follow-up consultations, periapical radiographs will be taken to check for the presence of periapical lesions.

REFERENCES:
- [Derived] Sobral APT, Santos EM, Leal Goncalves ML, Ferri EP, Junior WSB, Gimenez T, Gallo JMAS, Horliana ACRT, Motta LJ, Kalil Bussadori S. Efficacy of antibiotic and iodoform pastes in non-instrumental endodontic treatment of anterior primary teeth-Protocol for a randomized controlled clinical. PLoS One. 2023 Sep 8;18(9):e0291133. doi: 10.1371/journal.pone.0291133. eCollection 2023. PMID 37682887